CLINICAL TRIAL: NCT00276328
Title: Efficacy of Diosmectite (Smecta®) in the Treatment of Acute Diarrhoea in Adults. A Multicentre, Randomised, Double Blind, Placebo Controlled, Parallel Groups Study.
Brief Title: Study to Evaluate Smecta® vs Placebo on the Time to Recovery Following an Acute Diarrhoea Episode in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-31-00250-009
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Smectite; smecta

INTERVENTIONS:
Drug: Diosmectite (Smecta®)

SUMMARY:
The purpose of this study is to evaluate whether Smecta® is more effective than placebo with respect to time to recovery following an acute diarrhoea episode.

ELIGIBILITY:
Inclusion Criteria:

* Acute diarrhoea episode defined as at least 3 watery stools per day for 48 hours or less
* Patient with, usually, normal bowel habits, i.e. at least 3 stools per week and no more than 3 stools per day

Exclusion Criteria:

* Gross blood, pus in the stools
* Fever >39ºC
* Other episode of acute watery diarrhoea within the last 30 days
* History of chronic diarrhoea or motor diarrhoea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2005-01; Study Completion 2006-07

PRIMARY OUTCOMES:
Time to recovery ie time (hours) from the first sachet intake to the first formed stool (this formed stool must have been followed by a non-watery stool)

SECONDARY OUTCOMES:
Time (hours) from first sachet intake to the last watery stool
Number of stools and number of watery stools per 12 hour period
% of patients with recovery, per 12 hour period
% of patients with associated symptoms such as nausea, abdominal pain, anal irritation, per 12 hour period
Global evaluation of efficacy by the patient at Day 4 and Day 8 visits by a mean Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (31):
- Morocco (7):
  - Cabinet Médical, 50 rue Tata, Casablanca
  - Cabinet Medical, 17 Boulevard Bir Anzaran, Casablanca
  - Cabinet Médical, 12 rue Reaumur, Casablanca
  - Cabinet Médical, 94 boulevard du 11 janvier, Casablanca
  - Hopital Ibn Roched, Casablanca
  - Hôpital Ben Msick Sidi Othmane, Casablanca
  - Hôpital Avicenne, Rabat
- Tunisia (24):
  - Hopital régional de Ben Arous, Ben Arous
  - Hôpital des F.S.I., La Marsa
  - Hôpital Régional de Menzel, Menzel Bourguiba
  - Hôpital Fattouma Bourguiba, Monastir
  - Hôpital Régional, Nabeul
  - Hôpital Hédi Chaker, Sfax
  - avenue du 20 mars 1956 - Cité Jawhara, Sousse
  - Cité Laouina, Sousse
  - rue Abou Baker Essadik, Sousse
  - rue Alexandre Dumas, Sousse
  - rue Sidi Sahloul - Hammam, Sousse
  - rue Ali Ibn Taleb - Messadine, Sousse
  - Avenue Habib Bourguiba - Kalaa Essghira, Sousse
  - Avenue Habib Bourguiba - Sidi Bou Ali, Sousse
  - Cité Sahloul, route principale, AFH No.9, Sousse
  - Hôpital Sahloul, Sousse
  - rue du 1 er juin - Kalaa Kebira, Sousse
  - Polyclinique Taoufik, Tunis
  - Rue Micipsa, Tunis
  - Hôpital Charles Nicolle, Tunis
  - Hôpital La Rabta, Tunis
  - Hôpital Habib Thameur, Tunis
  - Hôpital Militaire, Tunis
  - Polyclinique de la CNSS, Tunis